CLINICAL TRIAL: NCT01170572
Title: Longitudinal Study of Vitamin D Metabolism and Bone Healing in Adult Patients With Recent Long Bone Fracture
Brief Title: Longitudinal Study of Patients Following Long Bone Fracture
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: London Deanery (Unknown)
Responsible Party: Sponsor
Other Study IDs: 007076; 10/H0805/6 (Other: REC number)
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Vitamin D; Long Bone Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Long bone fracture: Patients presenting to accident and emergency during the study period with long bone or clavicle fracture
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Studies in chickens show that blood levels of a particular form of vitamin D (called 24,25-dihydroxvitamin D) increase after bone fracture. Laboratory studies show that this form of vitamin D helps the bone healing process in chickens. The investigators want to find out whether blood levels of this form of vitamin D increase after bone fracture in humans. Previous research studies have not addressed this question. The results of this research could eventually lead to the development of new treatments to help bone healing after fracture.

Patients will be asked to take part in this study if they are aged 16 years or older and come to the Royal London Hospital with a broken bone in the arm or leg or collar bone (clavicle). They will be asked to give a 20ml (about 4 teaspoons) blood sample on three occasions: at the start of the study, at 5-14 days after the fracture; and at 4-10 weeks after the fracture. The rest of their normal care would not be affected. Follow-up blood samples will be timed to coincide with routine clinic visits which are scheduled as part of normal clinical care. Patients' vitamin D level will be measured as part of the study, and those who have a low vitamin D level will be informed about this, and advised about appropriate vitamin D supplementation. The investigators will let the patient or their GP know if any blood tests are abnormal

ELIGIBILITY:
Inclusion Criteria:

1. Any cross-shaft long bone or clavicle fracture within last 12 hours
2. Able to give written informed consent
3. Age ≥ 16 years
4. Fused physes (physiologically adult)

Exclusion Criteria:

1. Taking medication affecting vitamin D metabolism - carbamazepine, phenobarbital, phenytoin or primidone
2. Taking vitamin D supplement > 800 IU/day
3. Abdominal visceral injury, pleural injury (except pneumothorax), spinal cord injury, or GCS < 15 at presentation to hospital
4. Known Paget's disease, osteopetrosis, metastatic bone cancer, or primary bone cancer
5. Current prisoners
6. Currently taking part in another clinical research project

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the Accident and Emergency Department, Royal London Hospital, Whitechapel with a long bone or clavicle fracture
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Serum concentration of 24,25-dihyroxyvitamin D at 5-14 days post cross sectional long bone or clavicle fracture, compared with baseline. | 5-14 days post fracture

SECONDARY OUTCOMES:
Serum concentrations of vitamin D metabolites (including 1,25-dihydroxyvitamin D and 25-hydroxyvitamin D) and markers of bone healing | Baseline, 5-14 days, and 4-10 weeks post fracture
Peripheral blood expression of genes encoding enzymes in the vitamin D metabolic pathway. | Baseline, 5-14 days, and 4-10 weeks post fracture

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Martineau, MRCP, Study Director — Queen Mary University of London; Tim Harris, BM BS, Principal Investigator — Barts and the London NHS Trust
Locations (1):
- The Royal London Hospital, London, London, United Kingdom